CLINICAL TRIAL: NCT03413215
Title: Effects of Multidisciplinary Intensive Targeted Care in Improving Diabetes Outcomes: a Randomized Controlled Pilot Study - the Integrated Diabetes Education, Awareness and Lifestyle Modification in Singapore (IDEALS) Program
Brief Title: Effects of Multidisciplinary Intensive Targeted Care in Improving Diabetes Outcomes: a Pilot Study in Singapore
Acronym: IDEALS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changi General Hospital (Other)
Collaborators: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CGH-IDEALS
Record Dates: First submitted 2018-01-21; First posted 2018-01-29 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Diabetes Mellitus, Type 2; Diabetic Nephropathy; Hypertension
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Nephropathies; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): Patients randomized to the standard care group will receive usual care, which consists of clinic visits 4 monthly for review of BP, HbA1c and other investigations, and titration of medications;counseling with the diabetes nurse educator (DNE), and provision of educational materials on diabetes.
- Intensive (Experimental): Patient randomized to the intensive group will receive additional counselling and education by the DNE, medical social worker (MSW) on self-care and coping strategies for diabetes, and see the renal pharmacist for more intensive titration of antihypertensive medication between doctor visits. They will also be loaned blood pressure monitors and glucometers with test strips to perform self-monitoring at home in between outpatient visits. Smartphone and online technologies will be utilized to improve remote monitoring, education and self-care.
  Interventions: Behavioral: Intensive

INTERVENTIONS:
Behavioral: Intensive — Patients are provided with a BP machine, glucometer and test strips, and instructed how to use either a written or smartphone logbook, photograph their meals and use smartphone apps to measure daily activity. DNEs will contact patients in between visits to reinforce adherence and self-monitoring.
  MSWs will conduct at least 6 face-to-face sessions, at 3 weeks then less frequently, on essential self-care behaviours in people with diabetes: healthy eating; being physically active; monitoring of blood sugar; compliance with medications; problem-solving; healthy coping skills; and risk-reduction behaviour.
  Renal pharmacists will see patients at 2-4 week intervals for 3 months after the first clinic visit, and subsequently every 3-6 months. They will review patient's compliance, laboratory results and home BP, educate patient and titrate antihypertensives to meet BP goal. Physician referrals will be made for severe hypertension or hypotension, or intolerable side effects.
  Arms: Intensive

SUMMARY:
This study aims to investigate whether channeling purposefully structured resources to patients at high risk of developing diabetic complications to interdisciplinary team clinic consultations, interspersed with closer remote follow-up and aided by simple technology will be more effective than usual care in controlling diabetes mellitus, controlling multiple cardiovascular risk factors and reducing clinical event rates.

DETAILED DESCRIPTION:
The prevalence of diabetes in Singapore is estimated to grow from 400,000 to 670,000 by 2030 and an alarming one million by 2050 with the continuing rise in obesity prevalence. The current system currently has no formal stratification of patients for channelling of structured resources to patients that require more intensive treatment and follow-up (those at higher risk of progressing to having complications from diabetes due to poor glycemic control, or those who have signs of early complications).

We will therefore be researching effective health system delivery strategies to improve achievement of treatment targets (eg. HbA1c, blood pressure, LDL) and reduce vascular complications of diabetes mellitus (retinopathy, proteinuria, end stage renal disease, ischemic heart disease). These include:

* Stratification and channelling purposefully structured resources to patients with poorly controlled diabetes mellitus defined as having an HbA1c >9% on 2 or more occasions, and patients with diabetic complications (estimated glomerular filtration rate eGFR 30-60ml/min or proteinuria >0.5g/day or urine microalbumin:creatinine ratio >300mg/g)
* Training of all doctors/DNEs/dietitians involved in the counselling of patients in the field of motivational interviewing
* Providing easy accessibility to resources to allow patients to self-monitor their capillary blood glucose and blood pressure in between clinic visits - loaning of blood pressure units and glucometers for short (1-2 week) periods regularly
* Providing frequent telephone counselling by DNEs and Renal Pharmacists with regards to titration of medications, in particular ACE-inhibitors or angiotensin-receptor blockers to reach treatment targets
* Utilisation of social media and smart phone/tablet applications for relevant patients to improve and increase patient-healthcare professional interaction with regards to diabetes, provide daily bite-sized education via tablet/smart phone media/social media and improve compliance to exercise targets

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients aged 21-70 years
* Poorly controlled diabetes with microalbuminuria as defined by the following HbA1C > 9.0% with eGFR30- 60 ml/min and/or proteinuria >0.5g/day and/or urine microalbumin:creatinine ratio >300 mg/g on 2 consecutive measurements 3 months apart

Exclusion Criteria:

* Type 1 diabetes defined as a history of ketosis at diagnosis [acute symptoms with heavy ketonuria (>3+) or ketoacidosis] or continuous requirement of insulin within one year of diagnosis.
* Psychiatric conditions on medication
* On weight loss medications or have had bariatric surgery
* Life expectancy less than 12 months due to advanced cancers or other life-threatening conditions

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite primary endpoint | 3 years
  Composite of
  Incidence of all diabetes-related endpoints including:
  1. cardiovascular events (acute myocardial infarction, revascularisation procedures, heart failure, unstable angina, arrhythmia, stroke, transient ischemic attacks requiring hospital admissions) and related death
  2. chronic kidney disease (eGFR<60 ml/min/1.73m2) or end stage renal disease (dialysis and/or eGFR<15 ml/min/1.73m2) and related death
  3. visual impairment (corrected visual acuity of 20/200 or worse) or eye surgery (cataract removal, retinal surgery and vitrectomy)
  4. lower extremity amputation or foot ulcers requiring hospitalizations
  5. major infections - pulmonary and non-pulmonary requiring hospitalizations
  6. all-site cancers
  7. death

SECONDARY OUTCOMES:
Composite secondary endpoint | 3 years
  Proportions of patients with improved control of risk factors defined as:
  a) 2 or more of the 'ABC' targets: i) HbA1c<7% ii) BP<130/80 mmHg iii) LDL-C <2.6 mmol/L b) and/or c) 2 of the following changes in risk factor control: i) at least 0.5% reduction in HbA1c ii) at least 5 mmHg reduction in systolic BP iii) at least 0.5 mmol/L reduction in LDL-C iv) at least 3% reduction in body weight

CONTACTS AND LOCATIONS:
Overall Officials: Joan Khoo, FRCP, Principal Investigator — joan.khoo.j.c@singhealth.com.sg
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Phan TP, Alkema L, Tai ES, Tan KH, Yang Q, Lim WY, Teo YY, Cheng CY, Wang X, Wong TY, Chia KS, Cook AR. Forecasting the burden of type 2 diabetes in Singapore using a demographic epidemiological model of Singapore. BMJ Open Diabetes Res Care. 2014 Jun 11;2(1):e000012. doi: 10.1136/bmjdrc-2013-000012. eCollection 2014. PMID 25452860
- [Background] Shaw RJ, McDuffie JR, Hendrix CC, Edie A, Lindsey-Davis L, Nagi A, Kosinski AS, Williams JW Jr. Effects of nurse-managed protocols in the outpatient management of adults with chronic conditions: a systematic review and meta-analysis. Ann Intern Med. 2014 Jul 15;161(2):113-21. doi: 10.7326/M13-2567. PMID 25023250
- [Background] Chan JC, Gagliardino JJ, Baik SH, Chantelot JM, Ferreira SR, Hancu N, Ilkova H, Ramachandran A, Aschner P; IDMPS Investigators. Multifaceted determinants for achieving glycemic control: the International Diabetes Management Practice Study (IDMPS). Diabetes Care. 2009 Feb;32(2):227-33. doi: 10.2337/dc08-0435. Epub 2008 Nov 25. PMID 19033410
- [Background] Gaede P, Oellgaard J, Carstensen B, Rossing P, Lund-Andersen H, Parving HH, Pedersen O. Years of life gained by multifactorial intervention in patients with type 2 diabetes mellitus and microalbuminuria: 21 years follow-up on the Steno-2 randomised trial. Diabetologia. 2016 Nov;59(11):2298-2307. doi: 10.1007/s00125-016-4065-6. Epub 2016 Aug 16. PMID 27531506
- [Derived] Cashmore BA, Cooper TE, Evangelidis NM, Green SC, Lopez-Vargas P, Tunnicliffe DJ. Education programmes for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 Aug 22;8(8):CD007374. doi: 10.1002/14651858.CD007374.pub3. PMID 39171639
- [Derived] Tan E, Khoo J, Gani LU, Malakar RD, Tay TL, Tirukonda PS, Kam JW, Tin AS, Tang TY. Effect of multidisciplinary intensive targeted care in improving diabetes mellitus outcomes: a randomized controlled pilot study - the Integrated Diabetes Education, Awareness and Lifestyle modification in Singapore (IDEALS) Program. Trials. 2019 Sep 2;20(1):549. doi: 10.1186/s13063-019-3601-3. PMID 31477163